CLINICAL TRIAL: NCT05000970
Title: Telehealth Referral to Improve Outcomes for Asymptomatic Hypertension in the Emergency Department
Brief Title: Telehealth Referral to Improve Outcomes
Acronym: TRIO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AT&T and Vital Tech (Unknown)
Responsible Party: Principal Investigator, Kimberly T Souffront, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 20-01947
Record Dates: First submitted 2021-04-28; First posted 2021-08-11 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
Keywords: Asymptomatic hypertension; Referral; Telehealth; Remote patient monitoring; Emergency Department; blood pressure
MeSH Terms: conditions — Hypertension; Emergencies

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participant and investigator will be blinded on the study assignment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- TRIO PLUS tablet and nurse at day 3 (Experimental): Virtual nurse encounter at 3 days
  Interventions: Device: blood pressure cuff PLUS tablet; Other: Telehealth Consult
- TRIO PLUS Tablet and nurse at day 3 and 7 (Experimental): Virtual nurse encounter at 3 days and 7 days
  Interventions: Device: blood pressure cuff PLUS tablet; Other: Telehealth Consult
- TRIO PLUS Group (Placebo Comparator): No encounter
  Interventions: Device: blood pressure cuff PLUS tablet

INTERVENTIONS:
Device: blood pressure cuff PLUS tablet — all arms
  Other Names: wireless BP monitor and tablet
Other: Telehealth Consult — Telehealth consult with an RN
  Arms: TRIO PLUS Tablet and nurse at day 3 and 7; TRIO PLUS tablet and nurse at day 3

SUMMARY:
Emergency patients often have uncontrolled asymptomatic hypertension upon discharge from the emergency department. This 3-arm randomized controlled trial will evaluate the impact of nurse telehealth encounters and remote patient monitoring, using a software called Vital Tech, on blood pressure control and primary care engagement.

DETAILED DESCRIPTION:
Emergency Department (ED) clinicians encounter patients with asymptomatic hypertension (HTN) on a daily basis but usually fail to intervene. This pilot study will determine the utility of a novel intervention: Telehealth Referral to Improve Outcomes (TRIO), a conceptually driven information technology tool focused on patients who are asymptomatic and hypertensive upon ED discharge. It is designed to successfully link them to a primary care provider (PCP) after ED discharge to improve blood pressure (BP) control. 48 adult ED patients who have asymptomatic HTN (BP >/= 140/90 mmg and </= 180/120 mmHg) and who will be discharged will be enrolled in the study. This study is a single-site, 3-arm randomized controlled pilot trial. All patients will receive a wireless BP monitor and tablet. Group 2 (N=16) will additionally receive a telehealth consult with an RN at day 3. Group 3 (N=16) will additionally receive a telehealth consult with an RN at day 3 and day 7. The research team will collect feasibility outcomes: (recruitment rate, retention rate, and attrition rate of patients enrolled in TRIO at 6-months and 12-months. The research team will evaluate BP control and engagement with primary care at 6-months and 12-months and compare between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least two* high blood pressure readings during ED visit

  1. Systolic (top #) ≥140, ≤180 AND/OR
  2. Diastolic (bottom #) ≥ 90, ≤120

     *Second blood pressure may be confirmed when approaching the patient. Before approaching, check exclusions first.

     Exclusion Criteria:
* symptomatic hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  recruitment rate of patients enrolled in TRIO at 6-months.
Recruitment rate | 12 months
  recruitment rate of patients enrolled in TRIO at 12-months.
Retention rate | 6 months
  retention rate of patients enrolled in TRIO at 6-months.
Retention rate | 12 months
  retention rate of patients enrolled in TRIO at 12-months.
Attrition rate | 6 months
  attrition rate of patients enrolled in TRIO at 6-months.
Attrition rate | 12 months
  attrition rate of patients enrolled in TRIO at 12-months.

SECONDARY OUTCOMES:
Blood pressure | 6 months
Blood pressure | 12 months
Number of participant who had follow up care | 6 months
  Primary Care Engagement to be defined as having follow up care (yes/no) at 6 months
Number of participant who had follow up care | 12 months
  Primary Care Engagement to be defined as having follow up care (yes/no) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Souffront, PhD, APRN, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital Center Emergency Dept, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No